CLINICAL TRIAL: NCT00432731
Title: A Double-blind, Randomised, Controlled, Multi-centre Safety Study of a Refrigerator-stable Formulation of VARIVAX® in Healthy 12 to 15 Month-old Infants.
Brief Title: Safety Study of a Refrigerator-stable Formulation of VARIVAX®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: V210-061; X04-VAR-402 (Other: MCMVaccBV (SPMSD) Secondary ID)
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Varicella; Measles; Mumps; Rubella
Keywords: Prevention of : Varicella; Measles; Mumps; Rubella
MeSH Terms: conditions — Chickenpox; Measles; Mumps; Rubella | interventions — Chickenpox Vaccine

INTERVENTIONS:
Biological: VARIVAX®
Biological: M-M-RTM II

SUMMARY:
Primary objective:

To describe the safety profile of a refrigerator-stable formulation of VARIVAX® as a first single dose injection in 12 to 15 month-old infants in the 42-day follow-up period post-vaccination.

Secondary objectives: NA

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants from 12 months of age to 15 months of age.
2. Consent form signed by both parents or by the legal representative(s), properly informed about the study,
3. Parent(s) able to understand the protocol requirements and to fill in the Diary Card.

Exclusion Criteria:

1. Prior receipt of measles, mumps, rubella or varicella vaccine either alone or in combination vaccine,
2. Known or suspected clinical history of infection with measles, mumps, rubella, varicella or zoster,
3. Any known recent (≤30 days) exposure to measles, mumps or rubella,
4. Any known recent (≤30 days) exposure to varicella or zoster involving:
5. Any recent (≤3 days) history of febrile illness (rectal temperature ≥38.0°C),
6. Active untreated tuberculosis,
7. Any known blood dyscrasia, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems,
8. Any immune impairment or humoral/cellular deficiency, neoplastic disease or depressed immunity,
9. Any previous (≤150 days) receipt of immune serum globulin or any blood-derived products or scheduled to be administered through visit 3,
10. Any recent receipt of an inactivated or a live vaccine (≤ 30 days) or scheduled vaccination through visit 3

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500
Dates: Start 2004-12; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne FIQUET, MD, Study Director — SPMSD
Locations (25):
- France (24):
  - Amboise
  - Ancenis
  - Betton
  - Châteaubriant
  - Courbevoie
  - Essey-lès-Nancy
  - Floirac
  - Fougères
  - Garches
  - Gradignan
  - Issy-les-Moulineaux
  - Joué-les-Tours
  - Libourne
  - Lingolsheim
  - Mérignac
  - Nancy
  - Paris
  - Rueil-Malmaison
  - Strasbourg
  - Suresnes
  - Tours
  - Tresses
  - Vandœuvre-lès-Nancy
  - Villers-lès-Nancy
- Ragusa, Italy

REFERENCES:
- [Derived] Ferrera G, Gajdos V, Thomas S, Tran C, Fiquet A. Safety of a refrigerator-stable varicella vaccine (VARIVAX) in healthy 12- to 15-month-old children: A randomized, double-blind, cross-over study. Hum Vaccin. 2009 Jul;5(7):455-60. doi: 10.4161/hv.8269. Epub 2009 Jul 23. PMID 19305145